CLINICAL TRIAL: NCT07075250
Title: Safety and Efficacy of Realgar-Indigo Naturalis Formula（RIF） Combined With Anlotinib in the Treatment of Patients With Advanced Recurrent Platinum-Resistant Ovarian Cancer: A Prospective, Multicenter Clinical Study
Brief Title: Safety and Efficacy of RIF Combined With Anlotinib in the Treatment of Patients With Advanced Recurrent Platinum-Resistant Ovarian Cancer: A Prospective, Multicenter Clinical Study
Acronym: RIFOC003
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Peking University First Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tianjin People's Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Tianchang Yifan Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Xiaoping Li, Deputy Director, Institute of Obstetrics and Gynecology Research, Peking University People's Hospital, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHD008-001
Record Dates: First submitted 2025-06-25; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Platinum-resistant Ovarian Cancer (PROC)
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIF Combined with Anlotinib (Experimental)
  Interventions: Drug: Realgar-Indigo Naturalis Formulation Combined with Anlotinib

INTERVENTIONS:
Drug: Realgar-Indigo Naturalis Formulation Combined with Anlotinib — RIF: Oral administration after meals, 6 tablets each time, three times daily (tid), from day 1 to day 14 (d1-14), every 3 weeks (q3w), continuous dosing.
  Anlotinib : Oral administration before breakfast, 10 mg each time, once daily (qd), from day 1 to day 14 (d1-14), every 3 weeks (q3w), continuous dosing.
  Subjects will continue the study treatment until meeting the protocol-defined discontinuation criteria. The total treatment duration should not exceed 18 months.
  Other Names: anlotinib

SUMMARY:
This project plans to conduct a prospective, multicenter clinical study. The intended participants are patients with histologically confirmed advanced (FIGO III/IV stage) ovarian serous carcinoma, ovarian endometrioid carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma who have platinum-resistant recurrence or are platinum-refractory (n=30). The study design is a single-arm study. The treatment regimen for the study group is the RIF combined with anlotinib group, with continuous administration until disease progression, death, intolerable toxicity, loss to follow-up, withdrawal of informed consent, or study termination, whichever occurs first. The treatment duration will not exceed 18 months, with a follow-up period of 24 months.

The primary endpoint is progression-free survival (PFS). Secondary endpoints include overall survival (OS), objective response rate (ORR), disease control rate (DCR), quality of life score (QOL), and safety. The primary efficacy evaluation will use imaging methods (RECIST 1.1) combined with tumor marker CA125 levels.

All data in this study will be summarized using appropriate statistical measures based on data type: continuous data will be described using mean, standard deviation (STD), median, minimum, and maximum, while categorical data will be summarized using frequency and percentage (proportion). Time-to-event data will be analyzed using the Kaplan-Meier (KM) product-limit method to estimate median survival time, with survival curves plotted and 95% confidence intervals for median time estimated when necessary.

This study aims to evaluate the efficacy and safety of RIF combined with anlotinib in patients with platinum-resistant recurrent ovarian cancer, providing a new therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily participates in this study and signs the informed consent form.
2. Female aged 18-70 years.
3. Histologically confirmed advanced (FIGO stage III/IV) serous or ovarian endometrioid carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma.
4. Disease recurrence within 6 months after the last platinum-based chemotherapy or progression during chemotherapy (i.e., platinum-resistant or platinum-refractory).
5. ECOG performance status of 0 or 1, with an expected survival of ≥4 months.
6. Adequate organ function, meeting the following laboratory criteria within 14 days before enrollment:

   * **Complete blood count (without transfusion within 14 days):**

     1. Hemoglobin (Hb) ≥80 g/L;
     2. Absolute neutrophil count (ANC) ≥1.5×10⁹/L;
     3. Platelet count (PLT) ≥80×10⁹/L.
   * **Biochemical tests:**

     1. Total bilirubin ≤1.5×ULN (upper limit of normal);
     2. ALT and AST ≤2.5×ULN (≤5×ULN if liver metastases are present);
     3. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault formula).
   * **Cardiac function:** Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).
7. Ability to take oral medications.
8. ≥4 weeks since the last chemotherapy, radiotherapy, targeted therapy, immunotherapy, or other antitumor treatments before the first dose of study drugs.
9. Women of childbearing potential must agree to use highly effective contraception during the study and for 6 months after the last dose. A negative serum or urine pregnancy test within 7 days before enrollment is required, and the patient must be non-lactating.

Exclusion Criteria:

1. Prior treatment with arsenic agents (e.g., arsenic trioxide, Compound Huangdai Tablets) or anlotinib hydrochloride/other targeted therapies.

2. Known hypersensitivity to anlotinib or its excipients. 3. Known hypersensitivity to arsenic agents or their excipients. 4. **Comorbidities/medical history:**

1. Clinically significant hemoptysis (>50 mL/day within 3 months before enrollment) or active bleeding (e.g., gastrointestinal hemorrhage, hemorrhagic gastric ulcer, baseline fecal occult blood ≥++), or vasculitis.
2. Arterial/venous thromboembolic events within 6 months (e.g., cerebrovascular accident, deep vein thrombosis [unless catheter-related and resolved], pulmonary embolism).
3. Uncontrolled hypertension (systolic >140 mmHg or diastolic >90 mmHg despite medication) or history within 6 months of myocardial infarction, severe/unstable angina, NYHA class ≥2 heart failure, clinically significant arrhythmias, or symptomatic congestive heart failure.
4. Interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (e.g., pulmonary fibrosis, acute pneumonia).
5. Renal insufficiency: urine protein ≥++ or 24-hour urine protein ≥1.0 g.
6. Live attenuated vaccination within 28 days before the first dose or planned during the study.
7. HIV infection or AIDS; active hepatitis (HBV-DNA ≥500 IU/mL; HCV-RNA above detection limit) or coinfection with HBV/HCV.
8. Severe infection within 4 weeks (e.g., bacteremia, severe pneumonia requiring hospitalization) or active infection (CTCAE ≥grade 2) requiring systemic antibiotics within 2 weeks; unexplained fever >38.5°C during screening (unless tumor-related per investigator); active tuberculosis within 1 year.
9. Other malignancies within 3 years (except adequately treated basal cell carcinoma, squamous cell skin cancer, or cervical carcinoma in situ).
10. Palliative radiotherapy to >20% bone marrow within 1 week; history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
11. Major surgery within 28 days (diagnostic biopsies or PICC placement allowed).
12. Prior or planned allogeneic bone marrow or solid organ transplantation.
13. Peripheral neuropathy ≥grade 2; active brain metastases, leptomeningeal disease, or spinal cord compression (stable brain metastases treated ≥14 days before enrollment allowed if no hemorrhage on MRI/CT).

5. Current/recent (within 30 days) use of another investigational drug or participation in another clinical trial.

6. Conditions severely affecting oral drug absorption (e.g., dysphagia, chronic diarrhea, intestinal obstruction).

7. Any condition that may interfere with study results or compliance, per investigator judgment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS(Progression-Free Survival) | Evaluation at 3 months, 6 months, and 12 months of treatment

SECONDARY OUTCOMES:
OS(Overall Survival) | Evaluation at 3 months, 6 months, 12 months and 24 month of treatment
ORR(Objective Response Rate) | Evaluation at 3 months, 6 months, and 12 months of treatment
DCR((Disease Control Rate)) | Evaluation at 3 months, 6 months, and 12 months of treatment
QOL（Quality Of Life） | According to the EORTC QLQ-C30 criteria, evaluations were carried out at 3, 6, and 12 months of treatment.
  The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) is a widely used tool to assess the health-related quality of life (HRQoL) in cancer patients.
  1. Global Health Status/Quality of Life
     ≥70 points: Good quality of life (close to healthy population). 50-69 points: Moderate, with possible minor impact. <50 points: Poor, requiring clinical intervention.
  2. Functional Scales Physical Functioning (PF): Low scores indicate limitations in daily activities. Emotional Functioning (EF): Low scores suggest anxiety/depression risk, warranting psychological intervention.
     Social Functioning (SF): Low scores reflect negative disease impact on interpersonal relationships.
  3. Symptom Scales Fatigue (FA): Scores >50 indicate a need to evaluate anemia or treatment side effects.
  Pain (PA): Scores >40 require initiation of pain management. Nausea/Vomiting (NV): Scores >30 necessitate antiemetic regimen adjustment.
AE(Adverse Event) assessment | During the study up to 24 months

IPD SHARING:
Plan to Share IPD: No